CLINICAL TRIAL: NCT06527768
Title: The Effectiveness of a Theory-based Health Behaviour Change Intervention on Waist Circumference and Kidney Function in Patients of Metabolic Syndrome With Chronic Kidney Disease: A Pilot Randomised Controlled Trial
Brief Title: Theory-based Health Behaviour Change Intervention in Patients of Metabolic Syndrome With Chronic Kidney Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yan Linjia, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CERC Ref. No.: 2024.23.6
Record Dates: First submitted 2024-07-04; First posted 2024-07-30 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Diseases; Metabolic Syndrome
Keywords: Metabolic Syndrome; Chronic Kidney Disease; Waist Circumference; Kidney Function; Behaviour Change Intervention
MeSH Terms: conditions — Renal Insufficiency, Chronic; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theory-based health behaviour change intervention group (Experimental): Participants will be enrolled via WeChat and undergo 8 intervention sessions over 12 weeks. The 8 intervention sessions contain two online individual education sessions, two online group music-paced brisk walking training, two group discussions, and two telephone follow-ups. Besides, participants in the intervention group will be required to perform self-music-paced brisk walking 150 minutes/week for three months.
  Interventions: Behavioral: Theory-based health behaviour change interventio
- Control group (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Theory-based health behaviour change interventio — The online individual education sessions are related to MetS, CKD, healthy dietary and PA, displayed in the form of texts and pictures, and online instant conversations via WeChat. The online group music-paced brisk walking training includes a 5-minute warm-up, 30-minute music-paced brisk walking, and 5-minute stretching exercises to promote cool-down. The group discussion is related to current health status, recommended dietary regimens, and exercise and personal goals. The telephone follow-up after the group discussion is to reinforce the predetermined goals and the practice of healthy dietary and music-paced brisk walking, and to provide opportunities for answering any questions related to the practice of healthy dietary and music-paced brisk walking. All the education session contents are based on a well-structured health handbook. The self-music-paced brisk walking is required to be performed for 30 minutes/day, 5 days/week.
  Arms: Theory-based health behaviour change intervention group

SUMMARY:
The pilot study will adopt a 2-arm, pretest-posttest, and assessor-blind randomized controlled trial design to examine the feasibility and acceptability of a theory-based health behaviour change intervention and examine its effects on waist circumference (primary outcome), kidney function (estimated glomerular filtration rate, urine albumin-to-creatinine ratio, primary outcome), dietary behaviour, physical activity, exercise capacity and self-efficacy of diet behaviour and physical activity among Chinese adults with metabolic syndrome and chronic kidney disease.

Researchers will compare the theory-based health behaviour change intervention to usual care to see if the theory-based health behaviour change intervention can reduce waist circumference and preserve kidney function over three months.

A total of 40 adults with metabolic syndrome and chronic kidney disease will be recruited, with 20 participants in each group. Data will be collected at two-time points (baseline and immediate post-intervention) via an online questionnaire survey platform (Qualtrics) by researchers blinded to the group allocation to reduce the detection bias.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS) is a worldwide chronic disease mainly due to unhealthy diets and sedentary lifestyles. According to the International Diabetes Federation (IDF) definition of MetS, patients must have central obesity defined by waist circumference (WC) with ethnicity-specific values, plus any two of four additional factors, namely high triglycerides (TG), low high-density lipoprotein cholesterol (HDL-C), high fasting glucose (FG), and high blood pressure (BP).

More recent evidence indicates that the MetS could be an independent risk factor for chronic kidney disease (CKD). CKD is a progressive and incurable condition with high morbidity and mortality, which manifests as an estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 or a urine albumin-to-creatinine ratio (UACR) ≥ 30 mg/g for at least three months. According to KDIGO 2012 clinical practice guideline, CKD is divided into five stages (stages 1, 2, 3a, 3b, 4, 5), which are based on the eGFR test result, as the stage progresses, kidney function becomes more severe, ultimately leading to kidney failure. Previous studies have found that individuals with MetS had a higher risk of CKD compared with patients without MetS.

Central obesity, as the core component of MetS, could be one of the most essential pathogenes explaining the association between MetS and CKD. Central obesity mainly manifests as excess abdominal adipose tissue, which directly leads to the deranged synthesis of various adipose tissue cytokines (e.g., leptin, adiponectin, resistin, and visfatin) with nephrotoxic potential to cause sustained damage or structural changes to the kidneys, as well as indirectly trigger insulin resistance, dyslipidemia and hypertension, which are the most substantial risk factors for CKD.

Many patients fail to take MetS seriously until they are diagnosed with CKD. This is attributed to the additional complications and complex treatments associated with CKD, significantly affecting their daily lives. Current therapeutic guidelines for MetS suggest that non-pharmacological interventions (NPIs) with multifactorial lifestyle changes should be the primary treatment, including dietary modification, physical activity (PA), counselling or lifestyle modifications. Therefore, NPIs could be an essential method for reducing WC and preserving kidney function for the target population. Hence, this proposed study aims to develop an NPI for adults with MetS and CKD on the synthesized scientific evidence, and the effects on health-related outcomes will be evaluated using a randomized controlled trial (RCT) study.

Therefore, the design of the theory-based behavioural process change intervention is based on the findings of the systematic review (SR) and the implications of the qualitative study. Before the main RCT, a pilot RCT will be conducted to examine the feasibility and acceptability of the proposed intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants are 18 years old and above;
* Participants have both diagnoses of MetS based on IDF clinical diagnostic criteria (WC for Chinese: ≥ 90 cm in men and ≥ 80 cm in women, and fulfils two items of the following: TG ≥ 1.7 mmol/L or treatment for hypertriglycerides, HDL-C<1.03 mmol/L in men or <1.29 mmol/L in women or treatment for low HDL-C, FG ≥5.6 mmol/L or previously diagnosed type 2 diabetes, and BP ≥ 130/85 mmHg or treatment for hypertension). and CKD (eGFR < 60 mL/min/1.73 m2 or a UACR ≥ 30 mg/g for at least three months);
* No medical contraindications to exercise, including walking;
* Participants are capable of understanding and providing informed consent;
* Own a smartphone for accessing WeChat;
* Being able to communicate in Chinese;
* Stay in Chengdu during the study period.

Exclusion Criteria:

* Participants who cannot perform brisk walking exercise;
* Participants who have already started dialysis or kidney transplant;
* Current participation in another clinical trial related to health behaviour change or medical trial;
* Participants who have doctor-diagnosed psychiatric illness;
* Participants who have a cognitive impairment, which will be screened by the abbreviated mental test with a score lower than seven;
* Adjustment of medication within half a year;
* Participants who have performed regular planned exercise (Defined as at least 150 minutes of moderate-intensity aerobic activity or 75 minutes of high-intensity aerobic activity per week, or a combination of moderate-intensity and high-intensity aerobic activity) within the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Waist circumference | Data will be collected at day 0 and month 3.
  WC will be measured at the midpoint between the lower rib and the top of the iliac crest with the relaxed abdomen using a non-stretchable plastic measuring tape with an accuracy of 0.1 cm.
Estimated glomerular filtration rate | Data will be collected at day 0 and month 3.
  Blood samples will be obtained in the morning after fasting for at least 12 hours, and they will be refrigerated immediately after phlebotomy and centrifuged within 2 hours of collection. Blood samples will be analysed for eGFR. The eGFR will be calculated by the Chronic Kidney Disease Epidemiology Collaboration equation for Chinese individuals.
Urine albumin-to-creatinine ratio | Data will be collected at day 0 and month 3.
  Morning urine samples will be collected and refrigerated immediately to measure the levels of urine albumin and creatinine; then, the UACR will be calculated.

SECONDARY OUTCOMES:
Physical activity | Data will be collected at day 0 and month 3.
  The Chinese version of the short form of the International Physical Activity Questionnaire (IPAQ-SF) will be used to evaluate the amount of weekly PA. The IPAQ-SF records PA with nine questions, including vigorous, moderate-intensity, walking, and sitting. The simplified Chinese version of IPAQ-SF records self-reported physical activity in the last seven days, and the responses were converted to Metabolic Equivalent Task minutes per week (MET-min/wk). Total minutes over the last seven days spent on vigorous activity, moderate-intensity activity, and walking were multiplied by 8.0, 4.0, and 3.3, respectively, to create MET scores for each activity level.
Exercise capacity | Data will be collected at day 0 and month 3.
  The Six-Minute Walk Test (6MWT) will be used to evaluate exercise capacity. Participants will be asked to walk back and forth for six minutes at their usual speed along a straight 30-meter hospital corridor with marks every five meters. Throughout the test, participants will be permitted to slow down, pause, or take breaks as needed, but also be expected to resume walking when they feel ready. Encourage participants to use standard phrases from the guide. The 10-point Borg scale will be used to grade dyspnea and fatigue during the walk, with a higher score indicating a worse situation. The pulse oximeter will be used to measure heart rate and oxygen saturation, and the electronic sphygmomanometer will be used to measure blood pressure before and after the 6MWT. Additionally, the total distance covered will also be recorded.
Dietary behaviour | Data will be collected at day 0 and month 3.
  The diet control subscale of the Chinese version of Chronic Kidney Disease Self-care (CKDSC-DC) will used to measure the dietary behaviour. The CKDSC-DC is a 4-item scale that evaluates CKD-specific dietary self-care, with responses ranging from 1 (almost never) to 5 (almost always). Higher scores indicate better dietary self-management, and a total score of 14 or more is considered healthy.
Dietary behaviour | Data will be collected at day 0 and month 3.
  The nutrition domain of Health Promoting Lifestyle Profile-II (HPLP-II-N) will also be used to measure the dietary behaviour. The HPLP-II-N is a 9-item scale that assesses overall healthy dietary practices, with participants rating items on a 4-point scale from 1 (not at all) to 4 (always). A total HPLP-II-N score of 22.5 or greater is deemed healthy dietary behavior.
  Using both the CKDSC-DC and HPLP-II-N provides a comprehensive understanding of dietary behaviors among individuals with MetS and CKD. The CKDSC-DC offers a disease-specific measure of dietary self-care in CKD, while the HPLP-II-N evaluates broader aspects of health-promoting nutrition.
Self-efficacy of dietary behavior and physical activity | Data will be collected at day 0 and month 3.
  The Chinese version of the Health-Related Diet and Exercise Self-Efficacy Scale - Simplified Version (HRDESES) will be used to evaluate the self-efficacy of dietary behavior and physical activity. Response options are rated on a 5-point scale: zero (I'm not sure), one (mostly I cannot), two (I don't know), three (mostly I can), or four (I'm sure I can). The total score of HRDESES ranges from zero to 32, with a higher score indicating higher levels of health-related diet and exercise self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT06527768/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT06527768/ICF_001.pdf